CLINICAL TRIAL: NCT02140918
Title: Hemodynamic and Biological Effects of 3 Increasing Doses of Fludrocortisone in Healthy Volunteers
Brief Title: Fludrocortisone in Healthy Volunteers (AFLUCO4)
Acronym: AFLUCO4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013-004794-27
Record Dates: First submitted 2014-05-12; First posted 2014-05-16 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: Fludrocortisone; Mineralocorticoids; Hemodynamics; Pharmacokinetics
MeSH Terms: interventions — Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fludrocortisone 100 μg (Experimental): * 100 μg/day (25 µg four times daily) of fludrocortisone during 5 days
  * Investigations the sixth day
  Interventions: Drug: Fludrocortisone 100 μg
- Fludrocortisone 200 μg (Experimental): * 200 μg/day (50 µg four times daily) of fludrocortisone during 5 days
  * Investigations the sixth day
  Interventions: Drug: Fludrocortisone 200 μg
- Fludrocortisone 400 μg (Experimental): * 400 μg/day (100 µg four times daily) of fludrocortisone during 5 days
  * Investigations the sixth day
  Interventions: Drug: Fludrocortisone 400 μg
- Placebo (Placebo Comparator): * Placebo (four times daily) during 5 days
  * Investigations the sixth day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fludrocortisone 100 μg — Fludrocortisone 100 μg/day
  Arms: Fludrocortisone 100 μg
Drug: Fludrocortisone 200 μg — Fludrocortisone 200 μg/day
  Arms: Fludrocortisone 200 μg
Drug: Fludrocortisone 400 μg — Fludrocortisone 400 μg/day
  Arms: Fludrocortisone 400 μg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Fludrocortisone, in association with hydrocortisone, has demonstrated an improvement in survival in septic shock patients with relative adrenal insufficiency. However, the utility of low doses of steroids and in particular of mineralocorticoids in septic shock is still discussed.

The purpose of the investigators study is to investigate the effects of 3 increasing doses of fludrocortisone (100 μg, 200 μg, 400 μg) in order to determine which dose allows the best pressor response to phenylephrine in healthy volunteers, and simultaneously assess their respective hemodynamic and biological effects.

DETAILED DESCRIPTION:
In a previous study (AFLUCO2) in healthy volunteers with saline-induced hypoaldosteronism, the investigators found that single doses of both hydrocortisone and fludrocortisone induced a significant decrease in the pressor response to phenylephrine, probably due to a rapid non-genomic vasodilatory mechanism, and that these effects were additive.

The investigators also showed that, at the doses used in septic shock, hydrocortisone induced more pronounced mineralocorticoid effects than fludrocortisone and also induced systemic hemodynamic effects whereas fludrocortisone did not.

The investigators now want to perform a dose-response study under normal conditions (ie without saline-induced hypoaldosteronism) and after repeated administrations, to determine the optimal dose of fludrocortisone that allows an increase in the pressor response to phenylephrine and to characterize its concomitant hemodynamic and biological effects.

This placebo-controlled, randomized, double-blind, cross-over, 4-periods (fludrocortisone 100 μg/day, 200 μg/day, 400 μg/day, or placebo) study aims to investigate hemodynamic and biological effects of fludrocortisone administered orally during 5 days, in healthy volunteers.

Each period will be separated from the next one by a washout interval of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 25 years
* Body Mass Index between 20 kg/m² and 25 kg/m²
* Nonsmoker since at least 6 months
* Normal clinical examination, electrocardiogram and transthoracic echocardiography
* Normal routine biological parameters
* Written informed consent

Exclusion Criteria:

* History of significant allergy
* Resting heart rate < 50 bpm
* Subjects with abnormal hepatic or renal function, or cardiovascular, pulmonary, endocrine or psychiatric disease
* Ongoing medication during the study
* Alcohol consumption more than 30g/day or drug addiction
* Exclusion period mentioned on the national registry for clinical trials volunteers.
* Subject under legal protection

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Phenylephrine mean blood pressor dose-response relationship. | 1.5 hour after fludrocortisone administration

SECONDARY OUTCOMES:
Cardiac systolic and diastolic function assessed par transthoracic echocardiography during phenylephrine administration | between 1.5 and 2.5 hours after fludrocortisone administration
Systemic hemodynamic parameters | 30min before and 1h, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
  Systolic, diastolic and mean arterial pressures, heart rate, peripheral pulse pressure, cardiac output, stroke volume, systemic vascular resistances
Arterial stiffness : carotid-femoral pulse wave velocity | 30min before and 1h, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
Central aortic hemodynamic parameters | 30min before and 1h, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
  Aortic systolic, diastolic and mean arterial pressures, central pulse pressure, central pressure augmentation index (AIx)
Plasma parameters | 30min before and 1h, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
  Blood electrolytes, urea, creatinine, glucose, renin, aldosterone
Urinary parameters | 30min before and 2h, 4h, 6h after fludrocortisone administration
  Diuresis, urinary electrolytes, urea, creatinine, glucose
Area under the plasma concentration versus time curve (AUC) | Just before and 5min, 10min, 20min, 30min, 1h, 1h30, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
Plasma half-life of fludrocortisone | Just before and 5min, 10min, 20min, 30min, 1h, 1h30, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
Total Body Clearance | Just before and 5min, 10min, 20min, 30min, 1h, 1h30, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration
Apparent volume of distribution | Just before and 5min, 10min, 20min, 30min, 1h, 1h30, 2h, 3h, 4h, 5h, 6h after fludrocortisone administration

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD, Principal Investigator — Centre d'Investigation Clinique Inserm 1414, Service de Pharmacologie Clinique, Hôpital de Pontchaillou; Eric Bellissant, MD, PHD, Study Chair — Centre d'Investigation Clinique Inserm 1414, Service de Pharmacologie Clinique, Hôpital de Pontchaillou
Locations (1):
- Rennes University Hospital, Rennes, France